CLINICAL TRIAL: NCT03928158
Title: Sacubitril/Valsartan (LCZ696) in Patients With Advanced Hypertensive Left Ventricular Hypertrophy and Heart Failure With Preserved Ejection Fraction: Clinical, Haemodynamic and Neurohumoral Effects (a Phase 2, Randomized, Single-center, Parallel Group Study)
Brief Title: LCZ696 in Advanced LV Hypertrophy and HFpEF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Medical Research Center for Cardiology, Ministry of Health of Russian Federation (Other Government)
Responsible Party: Principal Investigator, Anastasiia Filatova, MD, PhD, principal investigator, MD, National Medical Research Center for Cardiology, Ministry of Health of Russian Federation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAA-A18-118022290061-2
Record Dates: First submitted 2019-04-23; First posted 2019-04-26 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure; Essential Hypertension
Keywords: left ventricular hypertrophy; diastolic dysfunction; LCZ696; HFpEF; HF; LV filling pressures
MeSH Terms: conditions — Heart Failure; Essential Hypertension; Hypertrophy, Left Ventricular | interventions — sacubitril and valsartan sodium hydrate drug combination; Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LCZ 696 (Experimental): Initial dose - 50 mg twice daily, up-titration to 200 mg twice daily. Patients will also receive standard therapy for heart failure (β-blockers, diuretics, MRAs)
  Interventions: Drug: LCZ 696
- Valsatran (Active Comparator): Initial dose - 40 mg twice daily, up-titration to 160 mg twice daily. Patients also will receive standard therapy for heart failure (β-blockers, diuretics, MRAs)
  Interventions: Drug: Valsartan

INTERVENTIONS:
Drug: LCZ 696 — 50-100-200 mg tablet
  Arms: LCZ 696
Drug: Valsartan — 40-80-160 mg tablet
  Arms: Valsatran

SUMMARY:
Patients with advanced LVH and HFpEF will be randomly assigned in open-label fashion to receive LCZ696 titrated to 200 mg twice daily or valsartan titrated to 160 mg twice daily, and will be treated for 24 weeks.

DETAILED DESCRIPTION:
Heart failure with preserved ejection fraction (HFpEF) has a signiﬁcant morbidity and mortality, and therapies that have proven effective in HF with reduced EF have not been shown to improve long-term prognosis in HFpEF. Inhibition of circulating neprilysin could augment deficient NP-receptor GC signaling and therefore be beneficial in HFpEF, as suggested by the decrease in NP following administration of valsartan/sacubitril in the phase 2 (PARAMOUNT study). Use of valsartan/sacubitril is currently being tested in the multicenter PARAGON-HF trial with HFpEF patients. The investigators suppose the best candidates for LCZ696 therapy will be patients with HFpEF and advanced concentric LV hypertrophy and obesity, i.e. having the lowest BNP bioavailability.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate/severe hypertensive left ventricular (LV) hypertrophy (LVMi ≥109 g/m² in women and ≥132 g/m² in men);
2. New York Heart Association (NYHA) class II-III heart failure;
3. Left ventricular ejection fraction > 50%;
4. Increased LV filling pressures assessed at rest or at peak exercise by echocardiography
5. Body mass index (BMI) > 30 kg/m²
6. Signed and data informed consent

Exclusion Criteria:

1. Age ≤ 18 years;
2. Evidence of myocardial ischemia during stress echocardiography;
3. Chronic atrial flutter or atrial fibrillation;
4. Alternative cause of left ventricular hypertrophy and impaired diastolic function (hypertrophic/restictive cardiomyopathy, aortic stenosis, constrictive pericarditis and etc.);
5. NYHA classification I or decompensated heart failure at screening;
6. Systolic blood pressure < 110 mmHg or > 180 mmHg;
7. Diastolic blood pressure < 40 mmHg or > 100 mmHg;
8. Anemia (Hb < 100 g/l);
9. Significant left sided structural valve disease;
10. Secondary hypertension;
11. Dyspnea due to non-cardiac causes such as pulmonary disease, anemia, severe obesity, primary valvular, or myocardial diseases;
12. Myocardial infarction or myocardial revascularization within the last 3 months of screening;
13. Stroke or TIA within the last 3 months of screening;
14. Autoimmunic and oncological diseases;
15. Impaired renal function, defined as eGFR < 30 ml/min/1.73 m²;
16. Impaired liver function;
17. Potassium concentration >5.2 mmol/L.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in 6-minute walking distance (6MWD) | 24 weeks
  Difference in distance walked during 6-minute walking test (6MWT) between 24 weeks after baseline and at baseline

SECONDARY OUTCOMES:
Change in exercise time during diastolic stress-test (DST) | 24 weeks
  Difference in exercise time during DST between 24 weeks after baseline and at baseline
Change in left atrial volume index (LAVI) | 24 weeks
  Difference in LAVI assessed by echocardiography between 24 weeks after baseline and at baseline
Change in average E/e' ratio | 24 weeks
  Difference in E/e' ratio assessed by echocardiography both at rest and at peak exercise during diastolic stress test (DST) between 24 weeks after baseline and at baseline
Change estimated pulmonary artery systolic pressure (PASP) | 24 weeks
  Difference in PASP assessed by echocardiography at peak exercise both at rest and at peak exercise during diastolic stress test (DST) between 24 weeks after baseline and at baseline
Change in left ventricular mass index (LVMI) | 24 weeks
  Difference in LVMI assessed by echocardiography between 24 weeks after baseline and at baseline
Change of New York Heart Association (NYHA) functional classification | 24 weeks
  Difference in NYHA class between 24 weeks after baseline and at baseline
Change in Minnesota Living With Heart Failure Questionnaire (MLHFQ) score | 24 weeks
  Difference in MLHFQ score between 24 weeks after baseline and at baseline. The questionnaire is comprised of 21 important physical, emotional and socioeconomic ways heart failure can adversely affect a patient's life. After receiving brief standardized instructions, the patient marks a 0 (zero) to 5 scale to indicate how much each itemized adverse of heart failure has prevented the patient from living as he or she wanted to live during the past 4 weeks. The questionnaire is simply scored by summation of all 21 responses. Score ranges from 0 (best quality of life) to 105 (worst quality of life).
Change in N-terminal pro b-type natriuretic peptide (NT-proBNP) | 24 weeks
  Difference in NT-proBNP plasma levels between 24 weeks after baseline and at baseline
Change in high-sensitivity C-reactive protein (hsCRP) | 24 weeks
  Difference in hsCRP plasma levels between 24 weeks after baseline and at baseline
Change in carboxyterminal propeptide of type I collagen (PICP) | 24 weeks
  DIfference in PICP plasma levels between 24 weeks after baseline and at baseline
Change in carboxyterminal telopeptide of type I collagen (CITP) | 24 weeks
  Difference in CITP plasma levels between 24 weeks after baseline and at baseline
Change in N-Propeptide Of Type III Procollagen (PIIINP) | 24 weeks
  Difference in PIIINP plasma levels between 24 weeks after baseline and at baseline
Change in Growth/differentiation factor 15 (GDF-15) | 24 weeks
  Difference in GDF-15 plasma levels between 24 weeks after baseline and at baseline
Change in sST2 | 24 weeks
  Difference in sST2 plasma levels between 24 weeks after baseline and at baseline
Change in Galectin-3 | 24 weeks
  Difference in Galectin-3 plasma levels between 24 weeks after baseline and at baseline
Change in monocyte chemoattractant-1 (MCP-1) | 24 weeks
  DIfference in MCP-1 plasma levels between 24 weeks after baseline and at baseline

CONTACTS AND LOCATIONS:
Locations (1):
- National Medical Research Center for Cardiology, Moscow, Russia